CLINICAL TRIAL: NCT05057364
Title: Heart Smart: A Virtual Self-Management Program for Homebound People With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sara Frye, MS OTR/L ATP, Therapy Professional Development Specialist, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 849646
Record Dates: First submitted 2021-08-31; First posted 2021-09-27 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: Heart failure; telehealth; occupational therapy; self-management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Pilot study, single group, no control. pre-post data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Smart Group (Experimental): Receives Heart Smart Intervention
  Interventions: Other: Heart Smart Virtual Self-Management Group

INTERVENTIONS:
Other: Heart Smart Virtual Self-Management Group — The Heart Smart Intervention is a 6 week virtual program consisting of one individual technology training session followed by 5 one hour group education sessions.

SUMMARY:
The purpose of this capstone project is to pilot Heart Smart, a virtual group program to improve self-efficacy for self-management skills for homebound people with heart failure.

DETAILED DESCRIPTION:
The purpose of this capstone project is to pilot Heart Smart, a virtual group program to improve self-efficacy for self-management skills for homebound people with heart failure. Heart Smart will provide synchronous virtual group education to homebound people with heart failure receiving services from Penn Medicine at Home. The primary clinical goal is to improve self-efficacy for heart failure self-management and improve their knowledge of heart failure self-management strategies. Secondary outcomes will explore the feasibility of the program by exploring technology, adherence and satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure
* Receiving home health care from Penn Medicine at Home at time of screening.
* Technology capabilities to participate in the program (laptop or tablet with a camera, internet access).
* Able to read and write in English.
* Cognitive ability to participate in the program if the participant is able to score12/15 on the Montreal Cognitive Assessment (MoCA) 5 Minute Phone Test.

Exclusion Criteria:

* Hearing impairment that impacts communication.
* Previous experience receiving occupational therapy services from the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Self-Efficacy Measure for Chronic Disease (SEMCD) | At first and final sessions (weeks 1 and 6)
  This self-report scale has 6 items which are each rated on a scale of 1 (not at all confident) to 10 (totally confident). The score for the scale is the mean of the scores for the six items. Possible scores are 1-10 with higher scores indicating higher self-efficacy. This scale is an appropriate outcome measure for a heart failure self-management group because it was designed to measure self-efficacy in people with chronic conditions such as heart failure and has undergone psychometric evaluation. This scale is free to use without permission. Administration takes less than 10 minutes.

SECONDARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) | At first and final sessions (weeks 1 and 6)
  This 23-item, Likert scale, self-report heart failure specific outcome measure. The instrument measures six domains: physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. This instrument is appropriate because it is designed for use for people with heart failure, will give an indication of participant heart failure severity for demographic purposes, and has a validated self-efficacy component. This scale requires a license which has been obtained for this pilot project. Administration takes less than 10 minutes. Scores range from 0 to 100 with higher scores indicating higher cardiac health status.
Change in Atlanta Heart Failure Knowledge Test V3 (AHFKT) | At first and final sessions (weeks 1 and 6)
  This 30 item multiple choice measure of heart failure self-management knowledge yields scores 0-30 which are commonly reported as a percentage (higher scores indicate more knowledge). Content validity was established through a panel of expert heart failure nurses.

OTHER OUTCOMES:
Attendance | At each weekly session for 6 weeks
  The number of participants at each meeting will be recorded.
Minutes of training | This will be recorded in the first session at week 1.
  The number of minutes spent in the pre-training session will be recorded.
Participant Satisfaction | At the final session on week 6
  Participants will answer three likert scale questions.
Technology failures | At each weekly session for 6 weeks.
  Total number of minutes missed per participant per session.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Frye, MS OTR/L ATP, Principal Investigator — Penn Medicine at Home Professional Development Department
Locations (1):
- Penn Medicine at Home, Bala-Cynwyd, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butler J, Khan MS, Mori C, Filippatos GS, Ponikowski P, Comin-Colet J, Roubert B, Spertus JA, Anker SD. Minimal clinically important difference in quality of life scores for patients with heart failure and reduced ejection fraction. Eur J Heart Fail. 2020 Jun;22(6):999-1005. doi: 10.1002/ejhf.1810. Epub 2020 Apr 2. PMID 32239794
- [Background] Butts B, Higgins M, Dunbar S, Reilly C. The Third Time's a Charm: Psychometric Testing and Update of the Atlanta Heart Failure Knowledge Test. J Cardiovasc Nurs. 2018 Jan/Feb;33(1):13-21. doi: 10.1097/JCN.0000000000000413. PMID 28481824
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014 Nov;67(11):1265-73. doi: 10.1016/j.jclinepi.2014.06.009. Epub 2014 Aug 3. PMID 25091546
- [Background] Spertus JA, Jones PG, Kim J, Globe D. Validity, reliability, and responsiveness of the Kansas City Cardiomyopathy Questionnaire in anemic heart failure patients. Qual Life Res. 2008 Mar;17(2):291-8. doi: 10.1007/s11136-007-9302-5. Epub 2007 Dec 29. PMID 18165909